CLINICAL TRIAL: NCT03060876
Title: Prospective Register Study of Patients After Proximal Humerus and Humerus Shaft Fracture for Data Collection of Healing Process, Quality of Life and Shoulder Function According to the Treatment Method - Hanover Humerus Register (HHR)
Brief Title: Hanover Humerus Registry
Acronym: HHR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Traumastiftung (Unknown)
Responsible Party: Sponsor
Other Study IDs: TS-1MHH2016-HHR
Record Dates: First submitted 2016-06-08; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2016-06

CONDITIONS: Proximal Humerus Fracture
Keywords: shoulder fractures; humeral fractures; operative therapy; conservative therapy; range of motion, articular; quality of life; proximal
MeSH Terms: conditions — Shoulder Fractures; Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This register study collects data of patients with proximal humerus and humerus shaft fractures to monitor the healing process by assessing shoulder function and quality of life according to the treatment method (operative or conservative management).

DETAILED DESCRIPTION:
This prospective data collection of patients with proximal humerus and humerus shaft fractures in a lifelong aftercare treatment plan is for analyzing the healing process in one patient and compared in the whole cohort.

According to actual scientific and clinical issues can this data collection be a basis in optimizing the treatment method.

ELIGIBILITY:
Inclusion Criteria:

* patients with trauma-related proximal humerus and humerus shaft fracture
* cognitively able to fill out a questionaire
* signed informed consent

Exclusion Criteria:

* patients with oncological-related proximal humerus and humerus shaft fracture
* cognitively not able to fill out a questionaire
* no informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with proximal humerus fracture
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Constant Shoulder Score (CS) (change over time) | following a aftercare treatment plan with follow ups after 6,12, 24, 52 weeks in the first year; then through study completion, an average of 1 year
  The CS is a commonly used outcome measure for assessing the outcomes of the treatment of shoulder disorders including the pain score, functional assessment, range of motion and strength measures.
  In week 6, 52 and in the yearly follow ups for comparison reasons the investigators also assess the CS of the not affected shoulder. Reported value is the impaired shoulder-functionality in percent. 100% are equivalent to an unimpaired shoulder function.
DASH (change over time) | following a aftercare treatment plan with follow ups after 1,3,6,12, 24, 52 weeks in the first year; then through study completion, an average of 1 year
  The Disabilities of the Arm, Shoulder and Hand (DASH) scoring system was developed to assess the level of disability for any patient with any condition affecting the upper limb by covering domains including symptoms, physical function, social function and psychological function.
Health related quality of life: EuroQoL (EQ-5D-3L+5L) (change over time) | following a aftercare treatment plan with follow ups after 1,3,6,12, 24, 52 weeks in the first year; then through study completion, an average of 1 year
  The EQ-5D-3L/5L is a standardized instrument for use as a measure of health outcome. It was designed for self-completion covering mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Furthermore, health state is indicated by a Visual Analog Scale (VAS). EQ-5D assesses the health status of the patients in an one-dimensional number (1-3/1-5).
Subjective Shoulder Value (SSV) (change over time) | following a aftercare treatment plan with follow ups after 1,3,6,12, 24, 52 weeks in the first year; then through study completion, an average of 1 year
  The SSV is defined as a patient's subjective shoulder assessment expressed as a percentage of an entirely normal shoulder, which would score 100%.

SECONDARY OUTCOMES:
healing process (change over time) | following a aftercare treatment plan with follow ups after 1, 3, 6,12, 24, 52 weeks in the first year; then through study completion, an average of 1 year
  Analyzing the radiological imaging for possible dislocation of fracture fragments or other complications
general health conditions | Baseline week 1
  Prior disorders of the affected shoulder and secondary diagnosis which are relevant for healing process of the proximal humerus fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Krettek, Prof. Doc., Principal Investigator — Hanover medical school trauma surgery// trauma foundation
Locations (1):
- Hanover medical school /trauma surgery, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Razaeian S, Hawi N, Zhang D, Liodakis E, Krettek C. Conservative treatment of displaced isolated proximal humerus greater tuberosity fractures: preliminary results of a prospective, CT-based registry study. Eur J Trauma Emerg Surg. 2022 Dec;48(6):4531-4543. doi: 10.1007/s00068-020-01453-7. Epub 2020 Sep 15. PMID 32930807